CLINICAL TRIAL: NCT01226693
Title: A Phase 1, Randomized, Open Label, Single Dose, 3 Treatment, Two Period, Balanced Incomplete Block Study In Healthy Fasted Volunteers To Assess The Safety, Tolerability, And Relative Oral Bioavailability Of A 6 Mg Dose Of The PH-797804 Material Sparing Tablet (MST) And Two Modified Versions Of The MST Formulation With And Without The Solubilizing Agent Sodium Lauryl Sulphate (SLS)
Brief Title: A Study In Healthy Volunteers To Assess The Safety, Tolerability, And Relative Oral Bioavailability Of Three Formulations Of PH-797804
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: A6631028
Record Dates: First submitted 2010-10-20; First posted 2010-10-22 (Estimated); Last update posted 2011-03-10 (Estimated); Status verified 2011-03

CONDITIONS: Healthy
Keywords: pharmacokinetic; single dose bioequivalence study; balanced incomplete block design; PH-797804; P38 kinase inhibitor
MeSH Terms: interventions — Sodium Dodecyl Sulfate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (6):
- Sequence 1 (Experimental)
  Interventions: Drug: PH-797804 material sparing tablet; Drug: PH-797804 Phase2b/3 with sodium lauryl sulphate
- Sequence 2 (Experimental)
  Interventions: Drug: PH-797804 Phase2b/3 with sodium lauryl sulphate; Drug: PH-797804 material sparing tablet
- Sequence 3 (Experimental)
  Interventions: Drug: PH-797804 material sparing tablet; Drug: PH-797804 Phase2b/3 without sodium lauryl sulphate
- Sequence 4 (Experimental)
  Interventions: Drug: PH-797804 Phase2b/3 without sodium lauryl sulphate; Drug: PH-797804 material sparing tablet
- Sequence 5 (Experimental): oral, 6mg, single dose
  Interventions: Drug: PH-797804 Phase2b/3 without sodium lauryl sulphate; Drug: PH-797804 Phase2b/3 with sodium lauryl sulphate
- Sequence 6 (Experimental): oral, 6mg, single dose
  Interventions: Drug: PH-797804 Phase2b/3 with sodium lauryl sulphate; Drug: PH-797804 Phase2b/3 without sodium lauryl sulphate

INTERVENTIONS:
Drug: PH-797804 material sparing tablet — oral, 6mg, single dose
  Arms: Sequence 1
Drug: PH-797804 Phase2b/3 with sodium lauryl sulphate — oral, 6mg, single dose
  Arms: Sequence 1
Drug: PH-797804 Phase2b/3 with sodium lauryl sulphate — oral, 6mg, single dose
  Arms: Sequence 2
Drug: PH-797804 material sparing tablet — oral, 6mg, single dose
  Arms: Sequence 2
Drug: PH-797804 material sparing tablet — oral, 6mg, single dose
  Arms: Sequence 3
Drug: PH-797804 Phase2b/3 without sodium lauryl sulphate — oral, 6mg, single dose
  Arms: Sequence 3
Drug: PH-797804 Phase2b/3 without sodium lauryl sulphate — oral, 6mg, single dose
  Arms: Sequence 4
Drug: PH-797804 material sparing tablet — oral, 6mg, single dose
  Arms: Sequence 4
Drug: PH-797804 Phase2b/3 without sodium lauryl sulphate — oral, 6mg, single dose
  Arms: Sequence 5
Drug: PH-797804 Phase2b/3 with sodium lauryl sulphate — oral, 6mg, single dose
  Arms: Sequence 5
Drug: PH-797804 Phase2b/3 with sodium lauryl sulphate — oral, 6mg, single dose
  Arms: Sequence 6
Drug: PH-797804 Phase2b/3 without sodium lauryl sulphate — oral, 6mg, single dose
  Arms: Sequence 6

SUMMARY:
There is no difference in the rate and extent of absorption of the material sparing tablet (MST), the Phase2b/3 formulation (P2b/3) with sodium lauryl sulphate (SLS) and the p2b/3 formulation without SLS.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and female subjects of non-childbearing potential between the ages of 21 and 55.
* No evidence of active or latent TB.
* An informed consent document signed and dated by the subject.

Exclusion Criteria:

* Evidence, including abnormal clinical laboratory parameters, eg, liver enzyme elevations, or a history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at time of dosing).
* Any condition possibly affecting drug absorption (eg, gastrectomy) or any active GI disease (including any relevant surgery).
* Any current and clinically significant skin lesions as described in Common Terminology Criteria for Adverse Events for Dermatology (CTCAE) Version 3. A clinically significant skin lesion is defined as Grade 1 (mild) for rash and pruritus, and Grade 2 (moderate) or above for all other lesions (see Short Name description in CTCAE for specific description of lesion).
* Use of prescription or nonprescription drugs, vitamins and dietary supplements within 7 days or 5 half-lives (whichever is longer) prior to the first dose of study medication.
* Other severe acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the subject inappropriate for entry into this study.

Ages: 21 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2010-11; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Area under the plasma concentration-time profile from time zero extrapolated to infinite time (AUCinf) | predose to day 7 of treatment period
Area under the plasma concentration-time profile from time zero to the time of the last quantifiable concentration (AUClast) | predose to day 7 of treatment period
Maximum observed concentration within the dosing interval (Cmax) | predose to day 7 of treatment period
Time for Cmax (Tmax) | predose to day 7 of treatment period
Terminal half-life (t1/2) | predose to day 7 of treatment period

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, Singapore, Singapore

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A6631028&StudyName=A%20Study%20In%20Healthy%20Volunteers%20To%20Assess%20The%20Safety%2C%20Tolerability%2C%20And%20Relative%20Oral%20Bioavailability%20Of%20Three%20Formulations%20Of%20PH-797804